CLINICAL TRIAL: NCT06586437
Title: Neuromodulation of the Cortex and Spinal Cord
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Father Flanagan's Boys' Home (Other)
Responsible Party: Principal Investigator, Max Kurz, Director of PoWER Lab, Father Flanagan's Boys' Home
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-25-XP
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Neuromodification; Brain; Spinal Cord; Upper Extremity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Cerebral Palsy participants will undergo baseline sham or stim intervention/brain imaging/clinical assessments, and then repeat with opposite intervention.
  Non-Cerebral Palsy controls will undergo the same baseline testing once as a reference group to determine a normative state of neuromodulation.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neurotypical Youth/Adults (Experimental): Compared with the sham controls, those receiving the transcutaneous current stimulation will demonstrate alterations in the strength of the sensorimotor cortical activity, spinal cord activity, and corticospinal coherence. Moreover, the extent of the alterations in the sensorimotor cortical activity, spinal cord activity, and corticospinal coherence will be tightly linked with the clinical presentations of persons with CP.
  Interventions: Behavioral: Clinical Assessments; Behavioral: Brain-Spinal Cord fMRI; Behavioral: Hoffmann Reflex Assessments; Behavioral: MEG Imaging; Behavioral: Transcutaneous Current Stimulation
- Cerebral Palsy Youth/Adults (Experimental): Compared with the sham controls, those receiving the transcutaneous current stimulation will demonstrate alterations in the strength of the sensorimotor cortical activity, spinal cord activity, and corticospinal coherence. Moreover, the extent of the alterations in the sensorimotor cortical activity, spinal cord activity, and corticospinal coherence will be tightly linked with the clinical presentations of controls.
  Interventions: Behavioral: Clinical Assessments; Behavioral: Brain-Spinal Cord fMRI; Behavioral: Hoffmann Reflex Assessments; Behavioral: MEG Imaging; Behavioral: Transcutaneous Current Stimulation

INTERVENTIONS:
Behavioral: Clinical Assessments — The participant will undergo a battery of clinical assessments to identify the upper extremity motor performance, sensory acuity, and ability to complete activities of daily living. Tests 1-5 will be completed separately for each hand. All participants will be video recorded while completing these assessments. The recordings will be used for grading tasks and data analysis: Box and Blocks, 9-hold peg board, Test of Arm Selective Control, Sensory Acuity Testing, KINARM End-Point Lab Sensory Test, Section GG of the inpatient Rehabilitaion Facility-Patient Assessment Instrument, NEURO-QOL Upper Extremity Function Scale, Edinburgh Handed Inventory
Behavioral: Brain-Spinal Cord fMRI — Resting state, brain-spinal cord activity, spinal cord microstructure, magnetic resonance spectroscopy
Behavioral: Hoffmann Reflex Assessments — Hmax 20-50 stimulations of increasing intensity. Next, the participant will sit quietly as 10 stimulations will be delivered at the participant's Hmax with an interstimulus interval of 15 seconds. Subsequently, stimulations at the participant's Hmax will be applied as the participants produce a contraction of 10-20% of their maximum voluntary contraction (MVC). The target contraction level will be shown in real-time based on the FCR EMG activity. The participant maintains their EMG activity at the target level for 6.5 seconds as 10 stimulations are delivered at the participants Hmax.
Behavioral: MEG Imaging — Resting state, somatosensory, isometric force matching, entrainment
Behavioral: Transcutaneous Current Stimulation — Cortical stimulation, spinal cord stimulation - sham and stim

SUMMARY:
Specific Aim 1: To further quantify the difference in the sensorimotor cortical activity, spinal cord activity, and corticospinal coherence of persons with CP.

Overall hypotheses: The sensorimotor cortical activity, spinal cord activity, and corticospinal coherence will be uncharacteristic in persons with CP when compared with neurotypical controls. Furthermore, the extent of the alterations in the sensorimotor cortical activity, spinal cord activity, and corticospinal coherence will be tightly linked with the clinical presentations of persons with CP.

Specific Aim 2: To investigate the effect of transcutaneous current stimulation applied over the cortex and/or spinal cord on the sensorimotor cortical activity, spinal cord dynamics, and corticospinal coherence.

Overall hypotheses: Compared with the sham controls, those receiving the transcutaneous current stimulation will demonstrate alterations in the strength of the sensorimotor cortical activity, spinal cord activity, and corticospinal coherence. Moreover, the extent of the alterations in the sensorimotor cortical activity, spinal cord activity, and corticospinal coherence will be tightly linked with the clinical presentations of persons with CP.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common pediatric motor disability, affecting 3.6 per 1000 children, and is typically a result of an insult to the developing brain. The brain insult impacts the precision of the motor actions and can have a lifelong impact on the precision of the motor actions. Although these motor deficits are vastly documented clinically, the underlying neurophysiological changes responsible for the emergence of these impairments are less understood. Our experimental work over the past decade has been directed at filling this knowledge gap. For example, magnetoencephalographic (MEG) brain imaging results were the first to show that the sensorimotor cortices of persons with CP exhibit abnormal activity when planning and executing a motor action, and that this aberrant activity is tightly coupled with slower reaction times and muscular force production errors. In addition, the investigators have repeatedly found that persons with CP have uncharacteristic activity within the somatosensory cortices following peripheral stimulation of the foot and hand, and that such abnormal cortical activity persists while producing a motor action. More recently, the investigators have evaluated if the altered cortical activity has cascading effects on the spinal cord interneuron dynamics. The logic for this premise was based on prior animal models that have shown that the initial insult to the developing brain impacts the structural organization of the spinal cord. The investigators' high-resolution structural MRI pipelines have revealed that the spinal cords of persons with CP have less grey and white matter area notable microstructural aberrations in the lemniscal and corticospinal tracts. Furthermore, the investigators' neurophysiological tests have indicated that persons with CP cannot excite the spinal cord's higher-threshold type II motor units that govern the fast-twitch fibers and the production of larger muscular forces. Altogether the investigators' body of experimental work suggests that there are unique interactions between the cortex and spinal cord that are likely responsible for the altered motor actions seen in those with CP. Further investigation of the brain and spinal cord connectivity will be important for advancing our understanding of the neurophysiology of persons with CP and the development of personalized therapeutic approaches that specifically target these deficiencies.

Transcutaneous current stimulation over the cortex and spinal cord is the most common noninvasive stimulation paradigms being explored with persons with CP in the hope of beneficially altering the neural generators that are involved in the production of a motor action. This approach involves the application of stimulating electrodes that emit a low-grade electrical current that passes through the skull/spine/skin to either excite or inhibit the underlying neural generators. The outcomes from these investigations have largely been mixed with some persons with CP demonstrating beneficial improvements, while others are non-responders. There are several limitations of these prior investigations. For one, there have been no neuroimaging investigations that have been performed to determine how the stimulation impacts the neurophysiology of the targeted cortical or spinal cord neural generators of those with CP. Secondarily, none of these prior investigations have considered whether these neuromodulation techniques impact the spinal cord-cortex connectivity. Lastly, many of the initial investigations have been case series that have not included a sham control group. This makes it difficult to discern if the clinical improvements seen in persons with CP after transcutaneous current stimulation are due to the physical therapy or physical therapy plus the neuromodulation.

There are large knowledge gaps in our understanding of how the respective transcutaneous current stimulation approaches influence the neurophysiology of persons with CP and if the stimulation protocols are beneficially altering the neurophysiology. The lion's share of the current research is blindly applying these neuromodulation techniques in hopes of having a beneficial improvement. There is a critical need to robustly evaluate the effect of these neuromodulation techniques on the neurophysiology of those with CP before the investigators are well prepared to launch a clinical trial. The Aims of this investigation are directed at beginning to fill this substantial knowledge gap.

ELIGIBILITY:
Inclusion Criteria:

* For Cerebral Palsy Participants:
* Gross Motor Function Classification score (GMFCS) levels between I-IV
* For Neurotypical Controls:
* No known atypical neurodevelopment (e.g. autism, Down Syndrome, ADHD, etc.)

Exclusion Criteria:

* For Cerebral Palsy Participants:
* Pregnancy
* Any condition that, in the opinion of the investigator, is a contraindication to participation
* The presence of any ferrous metal implant, including orthodonture, which may interfere with the MEG data acquisition and/or be an MRI safety concern
* No orthopedic surgery in the last 6 months or metal in their body that would preclude the use of an MRI
* For Neurotypical Controls:

Pregnancy

* Any condition that, in the opinion of the investigator, is a contraindication to participation
* The presence of any ferrous metal implant, including orthodonture, which may interfere with the MEG data acquisition and/or be an MRI safety concern
* No orthopedic surgery in the last 6 months or metal in their body that would preclude the use of an MRI

Ages: 11 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure-Clinical Assessment | 1 hour
  A stimulus intensity will be incrementally increased or decreased from 0.1 to 10 mA as the subject verbally reports their first sensation of the stimulus or perceived loss of the stimulus sensation. The ascending and descending perception tests will be repeated 3 times. The mean of the intensities will be used as the primary outcome variable.
  The KINARM robot will passively move the participant's hand-arm to various positions in the workspace as they hold the graspable robotic arm. The participant can see the position of their hand as a white dot in the virtual reality display. Once the robot returns home, the participant repeats the same movement that the robot performed. The difference between the final position of the hand when the robot passively moved the participant's arm and the final position when the participant actively moved their arm will be the primary outcome variable.
Primary Outcome Measure- fMRI | 1 hour
  1. Resting State: Functional brain imaging will be performed while the participant looks at a fixation cross for 5 minutes.
  2. Brain-Spinal Cord Activity: Functional imaging of the activity in the brain and spinal cord will be acquired concurrently while the participant performs a grip force target matching task. This task will consist of squeezing a force transducer with the hand to animate a box that ascends vertically based on the amount of force applied to the transducer. Target forces will be 10% and 30% of the participant's maximum grip force. The target forces will be randomized. The participant is instructed to match the target forces as quickly and as accurately as possible. The experiment will be conducted separately for the left and right hands and will take 10 minutes each to complete.
  3. Spinal Cord Microstructure: Structural images of the spinal cord will be acquired while the participant watches a move. The total scan time will be 20 minutes.
Primary Outcome Measure - Hoffman Reflex Assessments | 1 hour
  A percutaneous nerve stimulation will be used to determine the participant's maximal H-wave (Hmax) of the flexor carpi radialis muscle. This will be determined through 20-50 stimulations of increasing intensity. Next, the participant will sit quietly as 10 stimulations will be delivered at the participant's Hmax with an interstimulus interval of 15 seconds. Stimulations at the participant's Hmax will be applied as the participants produce a contraction of 10-20% of their maximum voluntary contraction. The participant will be instructed to maintain their EMG activity at the target level for 6.5 seconds as 10 stimulations are delivered at the participants Hmax. The ratio between the mean H-reflex amplitude in the Active Condition and the mean H-reflex amplitude in the Resting Condition will be used as the primary outcome variable. This task will be completed with the non-dominant hand, which will be determined from the clinical assessments.
Primary Outcome Measure - MEG Brain Imaging | 1 hour
  1. Resting state: The participants will sit quietly in the MEG with their eyes closed for 5 minutes.
  2. Somatosensory: An electric percutaneous stimulator will be used to deliver a low-level electrical stimulation to the median nerve at a level that is below the motor threshold (i.e., doesn't generate a twitch in the thumb).
  3. Isometric Force Matching: Participants will grasp a force transducer that will animate a box vertically to place it inside a target force box that represents 10 and 30% of their maximal grip force. The participants will be instructed to position and hold the animated box inside the target box for 300 ms until the target box disappears. The disappearance of the target box will signify when to stop the sustained force production.
  Tasks 2 & 3 will be completed with the non-dominant hand, which will be determined from the clinical assessments.
Primary Outcome Measure - Transcutaneous Current Stimulation | 30 minutes
  For participants receiving transcutaneous current stimulation over the spinal cord, one electrode will be placed over C6 while the other will be placed on the shoulder. Participants will be blinded to if they are in the sham or active group. While receiving the stimulation, the participants will practice opening and closing their less dominant hand for 20 minutes. The less dominant hand will be determined from the clinical assessments performed at the baseline time point. The participant will once again undergo the fMRI, MEG, or H-reflex protocol (which ever they completed for the baseline assessments) after completing the stimulation session. At the end of the transcutaneous current stimulation, the participant will complete a questionnaire regarding the sensations felt during stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Max J Kurz, PhD, Principal Investigator — Father Flanagan's Boys' Home
Locations (1):
- Boys Town National Research Hospital, Boys Town, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI and all of the investigators have made a commitment to publish, in a timely manner, all of the relevant scientific information that they will derive during this project. Deidentified data will be made available upon reasonable request to the Principal Investigator (Dr. Kurz).
Supporting Information: Study Protocol, CSR
Time Frame: Upon completion of study and data analysis
Access Criteria: Contact Dr. Kurz
URL: https://www.instituteforhumanneuroscience.org/power-lab